CLINICAL TRIAL: NCT07221162
Title: A Phase 1, Open-Label, Safety and Immunogenicity Trial of Boost-2867, an IgG-Fc-RBD Fusion Protein Next Generation SARS-CoV-2 Booster Vaccine, Via Intranasal and Intramuscular Routes in Previously Vaccinated Adults
Brief Title: A Safety and Immunogenicity Trial of Boost-2867 Vaccine, Via Intranasal and Intramuscular Routes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 25-1106
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10-21

CONDITIONS: COVID-19
Keywords: Boost-2867; coronavirus; COVID; Intramuscular; Intranasal; Next Generation Booster; Phase 1; Vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — ProMune; Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1 (Experimental): Participants will be administered 50 micrograms of Boost-2867 without adjuvant, intramuscularly (IM), to previously vaccinated healthy adults. 3 sentinel participants, less than 50 years old, will be enrolled for safety review before enrolling the remainder. N = 20.
  Interventions: Biological: Boost-2867; Other: Sodium Chloride, 0.9%
- Cohort 2 (Experimental): Participants will be administered 5 micrograms of Boost-2867 with Alhydrogel (R) and CpG 7909 adjuvants, intramuscularly (IM), to previously vaccinated healthy adults. 3 sentinel participants, less than 50 years old, will be enrolled for safety review before enrolling the remainder. N = 20.
  Interventions: Drug: Aluminum Hydroxide Suspension; Biological: Boost-2867; Biological: CpG 7909; Other: Sodium Chloride, 0.9%
- Cohort 3 (Experimental): Participants will be administered 15 micrograms of Boost-2867 with Alhydrogel(R) and CpG 7909 adjuvants, intramuscularly (IM), to previously vaccinated healthy adults. 3 sentinel participants, less than 50 years old, will be enrolled for safety review before enrolling the remainder. N = 20.
  Interventions: Drug: Aluminum Hydroxide Suspension; Biological: Boost-2867; Biological: CpG 7909; Other: Sodium Chloride, 0.9%
- Cohort 4 (Experimental): Participants will be administered 50 micrograms of Boost-2867 with Alhydrogel (R) and CpG 7909 adjuvants intramuscularly (IM) to previously vaccinated healthy adults. 3 sentinel participants, less than 50 years old, will be enrolled for safety review before enrolling the remainder. N = 20.
  Interventions: Drug: Aluminum Hydroxide Suspension; Biological: Boost-2867; Biological: CpG 7909; Other: Sodium Chloride, 0.9%
- Cohort 5 (Experimental): Participants will be administered 20 micrograms of Boost-2867 without adjuvant, intranasally (IN) to previously vaccinated healthy adults.3 sentinel participants, less than 50 years old, will be enrolled for safety review before enrolling the remainder. N = 20.
  Interventions: Biological: Boost-2867; Other: Sodium Chloride, 0.9%
- Cohort 6 (Experimental): Participants will be administered 50 micrograms of Boost-2867 without adjuvant intranasally (IN) to previously vaccinated healthy adults. 3 sentinel participants, less than 50 years old, will be enrolled for safety review before enrolling the remainder. N = 20.
  Interventions: Biological: Boost-2867; Other: Sodium Chloride, 0.9%
- Cohort 7 (Experimental): Participants will be administered 125 micrograms of Boost-2867 without adjuvant intranasally, to previously vaccinated healthy adults. 3 sentinel participants, less than 50 years old, will be enrolled for safety review before enrolling the remainder. N = 20.
  Interventions: Biological: Boost-2867; Other: Sodium Chloride, 0.9%

INTERVENTIONS:
Drug: Aluminum Hydroxide Suspension — Aluminum hydroxide adjuvant.
  Arms: Cohort 2; Cohort 3; Cohort 4
Biological: Boost-2867 — Boost-2867 is a recombinant ~50 kDa SARS-CoV-2 RBD (KP.2 variant) S1 subunit joined to a human IgG1 Fc, forming a ~100 kDa homodimer.
Biological: CpG 7909 — CPG 7909 is a synthetic oligodeoxynucleotide used as an adjuvant.
  Arms: Cohort 2; Cohort 3; Cohort 4
Other: Sodium Chloride, 0.9% — 0.9% Sodium Chloride Injection

SUMMARY:
This phase 1 clinical trial will evaluate the safety, reactogenicity, and immunogenicity of Boost-2867, given intramuscular (IM) with or without adjuvant or intranasal (IN) without adjuvant, as a booster dose to previously vaccinated healthy adults. Each of the six study sites will be assigned to enroll either only participants who will receive IM administration (3 sites) or only participants who will receive IN administration (3 sites); no site will administer both IM and IN study product administrations. Within the IM and IN Arms the cohorts will be sequentially enrolled. The study is designed as a non-randomized, open-label, dose-escalation clinical trial evaluating one dose level of Boost-2867 without adjuvant administered IM, three dose levels of Boost-2867 with adjuvant administered IM, and three dose levels of Boost-2867 without adjuvant administered IN. A sample size of 140 participants (20 participants per dose cohort) is anticipated. To evaluate for early safety signals for this first-in-human trial, study product administration of participants enrolled for IM administration and those enrolled for IN administration will proceed in a staged fashion. For Cohorts 1 (IM administration without adjuvant) and 5 (IN administration), which may be enrolled and dosed concurrently, 3 sentinel participants under 50 years of age will be enrolled in each Cohort over at least 2 days. For each of those Cohorts independently, a safety review of halting rules and clinical safety data through at least Day 8 will be conducted by the Protocol Safety Review Team (PSRT) prior to enrollment of the remainder of the cohort. Enrollment, dosing, and safety oversight for IM Cohorts 2, 3, and 4 will proceed in the same fashion as Cohort 1, except that sentinel enrollment need not be spaced over at least 2 days. Similarly, for IN Cohorts 6 and 7, enrollment and safety oversight will proceed in the same fashion as Cohort 5, except that sentinel enrollment need not be spaced over at least 2 days.

The primary objectives are: 1) To evaluate the safety and reactogenicity of a single IM injection of three different antigen dose levels (5, 15, and 50 microgram) of Boost-2867 with Alhydrogel (R) (alum) and CpG 7909 adjuvants, and a single injection of 50 microgram Boost-2867 without adjuvant, in previously vaccinated healthy adults. 2) To evaluate the safety and reactogenicity of a single IN administration of three different antigen dose levels (20, 50, and 125 microgram) of Boost-2867 without adjuvant in previously vaccinated healthy adults.

DETAILED DESCRIPTION:
This phase 1 clinical trial will evaluate the safety, reactogenicity, and immunogenicity of Boost-2867, given intramuscular (IM) with or without adjuvant or intranasal (IN) without adjuvant, as a booster dose to previously vaccinated healthy adults. Each of the six study sites will be assigned to enroll either only participants who will receive IM administration (3 sites) or only participants who will receive IN administration (3 sites); no site will administer both IM and IN study product administrations. Within the IM and IN Arms the cohorts will be sequentially enrolled. The study is designed as a non-randomized, open-label, dose-escalation clinical trial evaluating one dose level of Boost-2867 without adjuvant administered IM, three dose levels of Boost-2867 with adjuvant administered IM, and three dose levels of Boost-2867 without adjuvant administered IN. A sample size of 140 participants (20 participants per dose cohort) is anticipated. To evaluate for early safety signals for this first-in-human trial, study product administration of participants enrolled for IM administration and those enrolled for IN administration will proceed in a staged fashion. For Cohorts 1 (IM administration without adjuvant) and 5 (IN administration), which may be enrolled and dosed concurrently, 3 sentinel participants under 50 years of age will be enrolled in each Cohort over at least 2 days. For each of those Cohorts independently, a safety review of halting rules and clinical safety data through at least Day 8 will be conducted by the Protocol Safety Review Team (PSRT) prior to enrollment of the remainder of the cohort. Enrollment, dosing, and safety oversight for IM Cohorts 2, 3, and 4 will proceed in the same fashion as Cohort 1, except that sentinel enrollment need not be spaced over at least 2 days. Similarly, for IN Cohorts 6 and 7, enrollment and safety oversight will proceed in the same fashion as Cohort 5, except that sentinel enrollment need not be spaced over at least 2 days. The primary objectives are: 1) To evaluate the safety and reactogenicity of a single IM injection of three different antigen dose levels (5, 15, and 50 microgram) of Boost-2867 with Alhydrogel (R) (alum) and CpG 7909 adjuvants, and a single injection of 50 microgram Boost-2867 without adjuvant, in previously vaccinated healthy adults. 2) To evaluate the safety and reactogenicity of a single IN administration of three different antigen dose levels (20, 50, and 125 microgram) of Boost-2867 without adjuvant in previously vaccinated healthy adults. The secondary objectives are: 1) To evaluate the systemic anti-Spike humoral immune responses of a single IM or IN administration of Boost-2867. 2) To evaluate nasal mucosal immunoglobulin A (IgA) and immunoglobulin G (IgG) responses after IM and IN administration.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent before initiation of any study procedures.
2. Able to understand and agree to comply with planned study procedures and be available for all study visits.
3. Non-pregnant adults, 18 through 64 years of age at the time of study product administration.
4. Participants of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception***.

   * These criteria apply to females who are in a heterosexual relationship who are of childbearing potential. Not of childbearing potential include post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, or tubal ligation/salpingectomy).

     * True abstinence is 100% of the time, no sexual intercourse (penis enters the vagina). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods.

       * Acceptable forms of primary contraception include a monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more before the participant's study product administration, intrauterine devices, birth control pills, and injectable/implantable/insertable/transdermal hormonal birth control products. Must have used at least one acceptable primary form of contraception for at least 30 days before study product administration and agree to continue at least one acceptable primary form of contraception through 60 days after study product administration.
5. Participants of childbearing potential must have a negative urine pregnancy test at screening and within 24 hours before study product administration.
6. In general good health*. *As determined by medical history and physical examination, including vital signs, to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of the safety of participants. Chronic medical diagnoses/ conditions should be stable for the last 30 days (i.e., no hospitalizations, ER, or urgent care for the condition). This includes no change in chronic prescription medication, dose, or frequency due to deterioration of the chronic medical diagnosis/condition 30 days before the study product administration. Any prescription change due to a change of health care provider, insurance company, etc., or done for financial reasons and in the same class of medication will not be considered a deviation of this inclusion criterion. Participants may be on chronic or as-needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity.
7. Receipt of a complete primary authorized or approved COVID-19 vaccine series and at least one booster*.

   * Booster may be either homologous or heterologous to the primary vaccine series. It must be an FDA-authorized/licensed vaccine, though doses may have been received during a clinical trial.
8. Clinical screening laboratory evaluations are within normal reference ranges or grade 1 with no clinical significance (NCS) per the investigator's discretion*.

   *White Blood Cells (WBCs) with differential, hemoglobin (Hgb), platelets (PLTs), Alanine Transaminase (ALT), Aspartate Transaminase (AST), Creatinine (Cr), Alkaline Phosphatase (ALP), Total Bilirubin (T. Bili). Alanine Transaminase (ALT), Aspartate Transaminase (AST), Alkaline Phosphatase (ALP), Total Bilirubin (T. Bili), and creatinine values below the reference range will not be exclusionary as these values below the reference range are clinically insignificant.
9. Must agree to have samples stored for secondary research.

Exclusion Criteria:

1. Positive SARS-CoV-2 PCR at screening.
2. Abnormal vital signs (Grade 1 or higher):

   *Grade 1 or higher is equivalent to: Systolic blood pressure (SBP) >/= 141 mmHg or </= 89 mmHg Diastolic blood pressure (DBP) >/= 91 mmHg Heart rate (HR) is >/= 101 beats per minute or </= 54 beats per minute Oral temperature >/= 38.0 degrees Celsius (100.4 degrees Fahrenheit)
3. Self-reported or medically documented SARS-CoV-2 infection (regardless of whether symptomatic or asymptomatic) within 16 weeks prior to study product administration.
4. Participant who is pregnant or breastfeeding.
5. Blood or plasma donation within 4 weeks before study product administration.
6. Receipt of antibody or blood-derived products within 90 days before study product administration.
7. Any self-reported or documented significant medical or psychiatric diseases* or any other condition that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation.

   *Significant medical or psychiatric conditions include but are not limited to drug or alcohol abuse within 6 months of enrollment, significant kidney disease, liver disease, ongoing malignancy, or recent diagnosis of malignancy in the last five years, excluding treated basal and squamous cell carcinoma of the skin and cervical carcinoma in situ, which are allowed.
8. Neurological or neurodevelopmental conditions*.

   *Including history of Bell's palsy, history of four or more migraine headaches in the past 12 months that interfered with normal daily activity or any migraine headache in the past 5 years that required emergency or inpatient medical care, epilepsy, seizures in the last 5 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease.
9. History of significant respiratory disease currently requiring daily medications, history of asthma in the past 5 years, or any treatment of respiratory disease exacerbations in the last 5 years.
10. History of cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), including any history of myocarditis, pericarditis, or uncontrolled cardiac arrhythmia.
11. Any autoimmune disease, including hypothyroidism, without a defined non-autoimmune cause.
12. Has an acute illness determined by the site PI or appropriate sub-investigator within 72 hours before study product administration*.

    *An acute illness that is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
13. Has a positive test result for hepatitis B surface antigen, hepatitis C virus RNA (by reflex testing), or human immunodeficiency virus (HIV) antigen/antibody test at screening.
14. Has any confirmed or suspected immunosuppressive or immunodeficient state such as asplenia, recurrent severe infections, and chronic* immunosuppressant medication within the past 6 months**.

    *Chronic means more than 14 continuous days.

    **Ophthalmic and topical steroids are allowed.
15. Has received any investigational study product within 60 days, or 5 half-lives, whichever is longer, before study product administration or is planning to receive one during the study.
16. Has a history of hypersensitivity or severe allergic reaction* to any previous licensed or unlicensed study products or the candidate study product components**.

    *(e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction)

    **See IB for study product formulation.
17. Received or plans to receive licensed inactivated/subunit vaccine within 14 days of study product administration or live vaccine within 28 days of study product administration.
18. Plan to receive a COVID-19 booster vaccine within the 180 days following study product administration.
19. Regular use of intranasal medications, including steroids, and sinus rinsing treatments*.

    *Participants must have had no intranasal medication use for 30 days before study product administration and do not plan to use intranasal medications for 30 days after study product administration for medications other than steroids and for 6 months after study product administration for intranasal steroids (including over-the-counter (OTC) fluticasone).Participants should not use nasal irrigation or sinus rinsing treatments (e.g., Neti pots or saline washes) for 28 days after the study product administration and 7 days before study visits for the duration of the trial.
20. Use of illicit intranasal drugs in the 5 years before study product administration or plans to use during the study.
21. Current smoker (including cigarettes, marijuana, and vaping) or smoking within the prior 3 months.
22. Planned international travel between product administration and Day 29 visit.
23. Any significant nasal or upper airway disease*. *Including, but not limited to, being prone to epistaxis, has a history of inflammatory rhinitis (including allergic rhinitis) that requires daily medications, cochlear implants, head/neck radiation history, anosmia/dysosmia, and certain ear, nose and throat (ENT) conditions, including major anatomic nasopharyngeal abnormality or sinus polyp disease due to chronic sinusitis.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
Occurrence of abnormal clinical safety laboratory adverse events. | Through day 8
Occurrence of adverse events of special interest (AESIs). | Through 6 months
Occurrence of medically attended adverse events (MAAEs). | Through 6 months
Occurrence of new onset chronic medical conditions (NOCMCs). | Through 6 months
Occurrence of Serious adverse events (SAEs). | Through 6 months
Occurrence of solicited local adverse events (AEs). | Through 7 days
Occurrence of solicited systemic adverse events (AEs). | Through 7 days
Occurrence of unsolicited adverse events (AEs) s. | Through 28 days

SECONDARY OUTCOMES:
Geometric mean (GM) of nasal mucosal anti-S binding Immunoglobulin A (IgA) antibodies. | Day 1 through 91
Geometric mean (GM) of nasal mucosal anti-S binding Immunoglobulin G (IgG) antibodies. | Day 1 through 91
Geometric mean (GM) of serum Anti-S Immunoglobulin A antibodies (IgA). | Days 1 through 181
Geometric mean fold rise (GMFR) from baseline of nasal mucosal anti-S binding Immunoglobulin A (IgA) antibodies. | Day 1 through 91
Geometric mean fold rise (GMFR) from baseline of nasal mucosal anti-S binding Immunoglobulin G (IgG) antibodies. | Day 1 through 91
Geometric mean fold rise (GMFR) from baseline of serum Anti-S Immunoglobulin A antibodies (IgA). | Days 1 through 181
Occurrence of serum Anti-S Immunoglobulin G (IgG) antibodies. | Days 1 through 181
Seroconversion rate | Days 1 through 181
  Where seroconversion is defined as at least a 4-fold increase in serum neutralizing antibody titers over baseline.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California San Francisco - Zuckerberg San Francisco General Hospital - Division of Human Immunodeficiency Virus, Infectious Disease, and Global Medicine, San Francisco, California
  - Center for Immunization Research, Johns Hopkins Bloomberg School Public Health, Baltimore, Maryland
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - University of Pittsburgh - Medicine - Infectious Diseases, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington